CLINICAL TRIAL: NCT05828498
Title: The Mediterranean Diet Contributes To The Treatment Of Bacterial Vaginitis
Brief Title: The Mediterranean Diet and Bacterial Vaginitis
Status: Completed | Type: Observational
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, AYBALA TAZEOGLU, assistant professor, Osmaniye Korkut Ata University
Other Study IDs: OsmaniyeKAUnaad
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Bacterial Vaginitis
Keywords: bacterial vaginitis; Mediterranean diet; treatment
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- grup 1: patients who were on a diet and had a Mediterranean Diet Adherence Scale ≥7 were included in the diet group
  Interventions: Dietary Supplement: THE Mediterranean diet
- grup 2: As the control group (group 2), 64 patients participated in the study.

INTERVENTIONS:
Dietary Supplement: THE Mediterranean diet — The Mediterranean diet was applied to the patients with bacterial vaginitis selected randomly. diet content and application techniques were explained to the patient.
  Groups: grup 1

SUMMARY:
This study aimed to determine the effect of the Mediterranean diet as medical nutrition therapy in addition to medical therapy in patients diagnosed with vaginitis.

DETAILED DESCRIPTION:
In the study, 256 patients were diagnosed with vaginitis in the Obstetrics and Gynecology clinic. BV was diagnosed in 189 (73.8%) of the patients. Twelve patients with a diagnosis of BV who did not want to participate were excluded from the study. The Mediterranean diet was recommended and explained to 113 of the remaining 177 patients. 49 (42.5%) patients were excluded because the Mediterranean Diet Adherence Scale was <7. 64 (57.5%) patients who were on a diet and had a Mediterranean Diet Adherence Scale ≥7 were included in the diet group (group 1) As the control group (group 2), 64 patients participated in the study.

A randomized controlled study was designed to investigate the effect of the Mediterranean diet on the treatment of vaginitis in patients diagnosed with BV and given medical treatment. The study was carried out with the collaboration of the Gynecology and Obstetrics Clinic and Diet Clinic.

Patients diagnosed with BV and given medical treatment were divided into two groups a diet group and a control group. Patients who were diagnosed with BV, given medical treatment, and recommended a Mediterranean diet, whose dietary compliance was controlled and compliant with the Mediterranean diet control questionnaire, who came to the control examination after two weeks and were accepted to participate in the study, were included in the diet group. Patients diagnosed with BV, given medical treatment, followed up two weeks later, and accepted to participate in the study were included in the control group. In the control examination, the patients were grouped and compared as responsive and resistant after treatment.

Data collection Demographic data (age, gender), anthropometric measurements, presence of comorbid disease, menopausal period, presence of diabetes mellitus (DM), medical history, an average of three-day food consumption, and results of vaginitis treatment in the control examination of the patients included in the study were recorded. In addition, the patient's birth history, delivery technique, vaginal operation history, and vaginitis history were questioned in her medical history.

Anthropometric measurements Body weight (kg), height (cm), total body and abdominal fat ratio of each patient were measured and recorded by the researcher. Body weights were measured by the dietitian using a standard weighing instrument sensitive to 100 g without shoes. Values were determined in kilograms. Height measurements were taken with a Harpenden Stadiometer without shoes, heels touching, feet open at 45º, arms hanging at attention, head in frankfort plane. Values were determined in centimeters. BMI was calculated with the formula of body weight/height squared. Total body and abdominal fat ratio were measured with Tanita. According to the international BMI classification of the World Health Organization; 30 kg/m² was classified as obese (17).

Nutrient consumption analysis The patients were asked to write a diary of the foods they consumed while coming to the control examination. In order for the diary of the foods records to be reliable, tea glass, water glass, bowl, dessert spoon, tablespoon, serving spoon, ladle, 1 slice of bread, 1 meatball measure of meat, chicken, fish, 1 slice of cheese and their quantities were shared visually. Detailed information was given with replica samples.The foods consumed daily were recorded in the Bebis program. The amount of energy received by the patients from the average daily food consumption (kcal/day), what percentage of the daily energy was obtained from carbohydrates (%), and daily protein and fiber consumption amount (gr) were calculated. The distribution of protein consumption amount as animals and vegetables was investigated. The frequency of daily consumption of vegetables, fruits, and grains was recorded.

Mediterranean diet compliance questionnaire The adherence to the Mediterranean diet of the patients in the diet group who came to the control examination was evaluated with the 'Mediterranean Diet Adherence Scale'. The scale includes the type of oil used by the participants in meals, daily olive oil consumption, fruit and vegetable portions, margarine-butter and red meat consumption, weekly wine, pulses, fish-sea products, nuts, pastry consumption, tomato sauce. olive oil and white meat instead of red meat. It consists of 14 questions about the choice, to which all points are added by taking 1 point or 0 points for each question asked according to the consumption amount of the participant (18). Patients with a Mediterranean Diet Adherence Scale score >7 were considered compliant with the diet and were included in the study.

Diagnosis and treatment of bacterial vaginitis The obstetrician and gynecologist made the diagnosis of BV. Vaginal culture and microbiological examination were applied by the physician when necessary. Oral or vaginal antibiotics (metronidazole, clindamycin) were administered according to the BV physician's preference.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with bacterial vaginitis and given medical treatment were divided into two groups as diet group and control group. Diagnosed with bacterial vaginitis, given medical treatment, not pregnant mediterranean diet recommended The patients whose diet compliance was controlled and complied with the Mediterranean diet control questionnaire, who came to the control examination after two weeks and were accepted to participate in the study were included in the diet group.

Exclusion Criteria:

* pregnant under 18 years old out of control Bacterial vaginitis patients who received 7 or less on the Mediterranean diet compliance scale and did not accept to participate in the study were excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — bacterial vaginitis is female disease
Study Population: It consists of non-pregnant women over the age of 18 who have been diagnosed with bacterial vaginitis.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
determine the effect of the Mediterranean diet in the treatment of vaginitis | up to 2 week
  Determining the response of bacterial vaginitis patients who follow the Mediterranean diet to the treatment according to the group that does not.

CONTACTS AND LOCATIONS:
Locations (1):
- Osmaniye Korkut ATA University, Osmaniye, Turkey (Türkiye)